CLINICAL TRIAL: NCT06916494
Title: A Single-Arm, Open-Label, Multicenter Pilot Study：Rutin Combined With Tislelizumab and GC (Gemcitabine and Cisplatin) for Platinum-refractory Muscle-Invasive Bladder Cancer
Brief Title: Pilot Study on Rutin Combined With Tislelizumab and GC (Gemcitabine and Cisplatin) as Neoadjuvant Therapy for Platinum-refractory Muscle-invasive Bladder Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xin Gou, Professor, First Affiliated Hospital of Chongqing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZZ2025-070-02
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-02

CONDITIONS: Muscle Invasive Bladder Cancer
MeSH Terms: interventions — Rutin; Gemcitabine; Cisplatin; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rutin combined with Tislelizumab and GC (Experimental): Patients with MIBC who exhibit no response (stable disease or progressive disease) after two cycles of neoadjuvant GC chemotherapy (Cisplatin 100 mg/m² D2 q3w and Gemcitabine 1000 mg/m² D1, D8 q3w) will receive two cycles of rutin (40 mg tid.) combined with tislelizumab (200 mg D1 q3w) and GC (Cisplatin 100 mg/m² D2 q3w and Gemcitabine 1000 mg/m² D1, D8 q3w). Safety and adversed events will be assessed after every cycle of combinational treatment. Therapeutic response will be evaluated by contrast-enhanced MRI, and surgical decisions (transurethral resection, partial cystectomy, or radical cystectomy) will be made by two senior urologists. Epigenetic alterations and changes in the immune microenvironment will be analyzed post-treatment.
  Interventions: Drug: Rutin; Drug: Gemcitabine, Cisplatin; Drug: Tislelizumab

INTERVENTIONS:
Drug: Rutin — Rutin 40 mg tid. Treatment will be given for 2 cycles (21 days per cycle)
Drug: Gemcitabine, Cisplatin — Cisplatin 100 mg/m² D2 q3w, and Gemcitabine 1000 mg/m² D1, D8 q3w. Treatment will be given for 2 cycles (21 days per cycle)
Drug: Tislelizumab — Tislelizumab 200 mg D1 q3w Treatment will be given for 2 cycles (21 days per cycle)

SUMMARY:
This trial aims to evaluate the efficacy, safety, and biological mechanisms of rutin combined with tislelizumab and GC(Gemcitabine and Cisplatin) in platinum-refractory muscle-invasive bladder cancer patients. Key research questions include:

1. Whether rutin regulates epigenetic mechanisms in tumor cells from platinum-refractory bladder cancer patients and modulates the tumor immune microenvironment.
2. Evaluating the safety and adverse events of the combination treatment in platinum-refractory bladder cancer patients.
3. Assessing the disease control rate in platinum-refractory bladder cancer patients receiving this therapy.

Patients with MIBC who exhibit no response (stable disease or progressive disease) after two cycles of neoadjuvant GC chemotherapy will receive two cycles of rutin combined with tislelizumab and GC. Safety and adverse events will be assessed after each cycle of combinational treatment. Therapeutic response will be evaluated by contrast-enhanced MRI, and surgical decisions (transurethral resection, partial cystectomy, or radical cystectomy) will be made by two senior urologists. Epigenetic alterations and the changes in immune microenvironment will be analyzed post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cT2-cT4N0M0 muscle-invasive bladder cancer (MIBC)
* No response after 2 cycles of GC neoadjuvant chemotherapy
* No prior use of systemic immunotherapy or target therapy
* Tumor is measurable according to New response evaluation criteria in solid tumours: Revised RECIST guideline
* ECOG (ZPS, 5-point scale) 0-1

Exclusion Criteria:

* Age less than 18 years
* Patients with severe cardiac, cerebral, hepatic, or renal disease
* Severely malnourished patients
* Patients with mental illness and those without insight and unable to express exactly
* Combined with malignant tumors of other organs
* Systemic infectious diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Tumor microenvironment | From enrollment to the end of treatment at 6 weeks
  Immune microenvironment and epigenetic alterations in bladder tumors, including immune cell components.

SECONDARY OUTCOMES:
Safety and adverse events | From enrollment to the end of treatment at 6 weeks
  The description of adverse events will be coded according to MedDRA terminology and graded according to NCI-CTCAE v5.0.
Objective remission rate | From enrollment to the end of treatment at 6 weeks
  The proportion of patients with complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD) after treatment was calculated according to established response evaluation criteria (Response Evaluation Criteria in Solid Tumors [RECIST], version 1.1).
  Definitions:
  CR (Complete Response): Disappearance of all target lesions with no new lesions.
  PR (Partial Response): ≥30% decrease in the sum of diameters of target lesions. SD (Stable Disease): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
  PD (Progressive Disease): ≥20% increase in the sum of diameters of target lesions and/or appearance of new lesions

CONTACTS AND LOCATIONS:
Overall Officials: Xin Gou, Professor, Study Chair — The First Affiliated Hospital of Chongqing Medica University
Locations (1):
- First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The study outcomes and follow-up information will be available after paper publication.
Supporting Information: Study Protocol, SAP
Time Frame: The IPD and supporting information will be available after 2027.12.31
Access Criteria: Study protocal of the study is available from professor Xin Gou (email:cymnk@163.com)